CLINICAL TRIAL: NCT01949129
Title: Allogeneic Stem Cell Transplantation for Children and Adolescents With Acute Lymphoblastic Leukaemia
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: St. Anna Kinderkrebsforschung (Other)
Collaborators: ALL SCTped Forum (Other); European Society for Blood and Marrow Transplantation (Network); ALL-BFM Study Group (Network); Assistance Publique - Hôpitaux de Paris (Other); Dutch Childhood Oncology Group (Other); Swiss Pediatric Oncology Group (Other); Australian & New Zealand Children's Haematology/Oncology Group (Other)
Responsible Party: Principal Investigator, Prof. Christina Peters, Univ.-Prof. Dr. Christina Peters, St. Anna Kinderspital, Austria
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALL SCTped FORUM 2012
Record Dates: First submitted 2013-09-09; First posted 2013-09-24 (Estimated); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Acute Lymphoblastic Leukaemia
Keywords: stem cell transplantation; children and adolescents; high risk acute lymphoblastic leukaemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Etoposide; Thiotepa; Acetyl-CoA C-Acyltransferase; treosulfan; fludarabine; Influenza Vaccines; Busulfan; thymoglobulin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Flu/Thio/Treo (Experimental): Fludarabine/Thiotepa/Treosulfan is used as conditioning regimen for haematopoietic stem cell transplantation (HSCT) in patients with:
  * MSD (matched sibling donors) or MD (matched related or unrelated donors). In addition, patients undergoing MD HSCT will receive ATG Thymo- or Grafalon.
  * MMD (mismatched donors) with CB (Cord blood) or TCD (T-Cell depletion) or CD34+ selection. In addition, these patients will receive ATG Thymo- or Grafalon.
  * MMD (mismatched donors) patients receiving Post TX-Cyclophosphamide
  Interventions: Drug: Thiotepa; Drug: Treosulfan; Drug: Fludarabine; Drug: ATG Thymoglobulin; Drug: Grafalon
- TBI/VP16 (Active Comparator): TBI (Total Body Irradiation) / VP16 is used as conditioning regimen for haematopoietic stem cell transplantation (HSCT) in patients older than 48 months with:
  * MSD (matched sibling donors) or MD (matched related or unrelated donors). In addition, patients undergoing MD HSCT will receive ATG Thymo- or Grafalon.
  * MMD (mismatched donors) with CB (Cord blood) or TCD (T-Cell depletion) or CD34+ selection. In addition, these patients will receive ATG Thymo- or Grafalon.
  * MMD (mismatched donors) patients receiving Post TX-Cyclophosphamide.
  Patients aged 24-48 months may optionally receive Total Body Irradiation (TBI).
  Interventions: Drug: VP16; Radiation: TBI; Drug: ATG Thymoglobulin; Drug: Grafalon
- Flu/Thio/ivBu (Experimental): Fludarabine/Thiotepa/iV Busulfan is used as conditioning regimen for haematopoietic stem cell transplantation (HSCT) in patients with:
  * MSD (matched sibling donors) or MD (matched related or unrelated donors). In addition, patients undergoing MD HSCT will receive ATG Thymo- or Grafalon.
  * MMD (mismatched donors) with CB (Cord blood) or TCD (T-Cell depletion) or CD34+ selection. In addition, these patients will receive ATG Thymo- or Grafalon.
  * MMD (mismatched donors) patients receiving Post TX-Cyclophosphamide
  Interventions: Drug: Thiotepa; Drug: Fludarabine; Drug: Busulfan; Drug: ATG Thymoglobulin; Drug: Cyclophosphamide; Drug: Grafalon
- Bu/VP16/Cy (Experimental): Busulfan/VP16/Cyclophosphamide is an alternative conditioning arm that may optionally be used for HSCT with MSD/MD and MMD graft in patients aged 0-24 months. Patients undergoing MD HSCT will also receive ATG Thymo- or Grafalon.
  Interventions: Drug: VP16; Drug: Busulfan; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: VP16 — 60 mg/kg BW,1 day in TBI/VP16 conditioning; 40 mg/kg BW in Bu/VP16/Cy conditioning
  Other Names: Etoposide
  Arms: Bu/VP16/Cy; TBI/VP16
Radiation: TBI — 2 x 2Gy/day , 3 days (total 12Gy)
  Arms: TBI/VP16
Drug: Thiotepa — 2x5 mg/kg BW, 1 day
  Other Names: Thio
  Arms: Flu/Thio/Treo; Flu/Thio/ivBu
Drug: Treosulfan — 14g/m² BS, 3 days
  Other Names: Treo
  Arms: Flu/Thio/Treo
Drug: Fludarabine — 30 mg/m² BS, 5 days
  Other Names: Flu
  Arms: Flu/Thio/Treo; Flu/Thio/ivBu
Drug: Busulfan — iV, dosage according therapeutic drug monitoring, 4 days
  Other Names: Bu
  Arms: Bu/VP16/Cy; Flu/Thio/ivBu
Drug: ATG Thymoglobulin — MD: ATG Thymo: 2,5mg/kg BW/d 3 days.
  Other Names: ATG Thymo
  Arms: Flu/Thio/Treo; Flu/Thio/ivBu; TBI/VP16
Drug: Cyclophosphamide — as part of conditioning 60 mg/kg BW 2 days or as GvHD Prophylaxis 50mg/kg BW/d 2 days with Mesna
  Other Names: Cy
  Arms: Bu/VP16/Cy; Flu/Thio/ivBu
Drug: Grafalon — MD: 15mg/kg BW/d 3 days MMD: 10mg/kg BW/d 3 days
  Other Names: Anti-human T-lymphocyte immunoglobulin
  Arms: Flu/Thio/Treo; Flu/Thio/ivBu; TBI/VP16

SUMMARY:
The ALL SCTped 2012 FORUM is a multinational, multi-centre, controlled, prospective phase III study for the therapy and therapy optimisation for children and adolescents with ALL in complete morphological remission (CR, less than 5% bone marrow blasts, no blasts in cerebrospinal fluid, no other extramedullary leukemia), who have an indication for HSCT with a myeloablative conditioning regimen.

The stratification of patients in first and following remissions according to the individual transplantation modalities rests upon an indication for allogeneic HSCT and the availability of a suitable donor within the individual transplantation groups.

DETAILED DESCRIPTION:
Acute and late side effects of TBI in combination with other chemotherapeutic are manifold to the growing organism and include severe organ dysfunction/failure due to toxicity. Although transplant associated mortality was reduced after HSCT in the last decade due to better HLA matching, infection prevention and control, the burden of late complications is still a matter of concern. Growth retardation, hormonal dysfunction, sterility and the risk of secondary cancer are the late consequences of TBI in children. However, so far no prospective study has demonstrated similar outcomes in paediatric ALL using chemo-conditioning regimen before HSCT. The reason for that is manifold: only a minority of children with ALL qualifies for allogeneic HSCT as most patients are cured with sole modern chemotherapy approaches. Those with dismal prognosis are treated in HSCT centres offering a care to patients with different diseases. Therefore it is nearly impossible to answer the complex outcome questions in single centres or even in single countries. International cooperation is essential to allow prospective investigation within comparable patient cohorts.

The trial was initiated to investigate whether chemotherapy based conditioning could replace TBI in pediatric patients with acute lymphoblastic leukemia (ALL) undergoing allogeneic hematopoietic stem cell transplantation (HSCT). It was registered and approved as a prospective, randomized, controlled, open-label, international, multicenter, phase III, non-inferiority trial. Pediatric patients with acute lymphoblastic leukemia (ALL) aged ≤18 years at diagnosis and 4-21 years at HSCT in complete remission pre-HSCT, and with an HLA-compatible related (MSD) or unrelated donor (MD) were randomly assigned to myeloablative conditioning with fractionated 12 Gy TBI and etoposide versus fludarabine (Flu), thiotepa (Thio), and either busulfan (Bu) or treosulfan (Treo). The decision to use the irradiation-free conditioning or Flu/Thio/Treo or Flu/Thio/ivBu was country specific. Patients aged < 4 years received irradiation-free conditioning. Patients with a mismatched donor (MMD) were stratified according to the donor's stem cell source (cordblood, haploidentical tx or bone marrow/peripheral blood stem cells).

The stopping rule was applied on March 31, 2019 following a suspension of random assignment in December 2018 after the chemoconditioning was proven to be significantly inferior to TBI. As a result, TBI/VP16 conditioning remains the standard for patients older than 4 years with MSD/MD, but the age limit for TBI/VP16-based conditioning may be optionally lowered to 2 years.The use of Flu/Thio/Treo or Flu/Thio/ivBu conditioning in this age group is made at centre level based on individual patient assessment. Alternatively, patients aged 0-2 years may receive Bu/VP16/Cy at the discretion of the treating physician.

The MSD/MD randomised patients remain in a follow-up to explore the impact of risk factors on the incidence of Adverse Events of Special Interest (AESIs) and on overall survival and event free survival in the entire MSD/MD cohort.

In MMD patients, event free survival (EFS) after HSCT from HLA mismatched donors using mismatched unrelated donors (MMD), mismatched cord blood or HLA haplo-identical family members is observed

ELIGIBILITY:
Inclusion Criteria:

Patients with ALL (except for patients with B-ALL) who fulfil the following criteria:

* age at diagnosis ≤ 18 years. Age at HSCT ≤ 21 years
* indication for allogeneic HSCT
* complete remission (CR) before HSCT
* written consent of the parents (legal guardian) and, if necessary, the minor patient via "Informed Consent Form"
* no pregnancy
* no secondary malignancy
* no previous HSCT
* HSCT is performed in a study participating centre

Exclusion Criteria:

* patients who do not fulfil the inclusion criteria
* Non Hodgkin-Lymphoma
* the whole protocol or essential parts are declined either by patient himself/herself or the respective legal guardian
* no consent is given for saving and propagation of anonymous medical data for study reasons
* severe concomitant disease that does not allow treatment according to the protocol at the investigator's discretion (e.g. malformation syndromes, cardiac malformations, metabolic disorders)
* Karnofsky / Lansky score < 50%
* subjects unwilling or unable to comply with the study procedures

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1800 (Estimated)
Dates: Start 2013-04; Primary Completion 2025-06 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) Stratum 1a (randomisation TBI+ chemo-conditioning vs. chemo-conditioning only) | first: 18 months after inclusion of first patient, afterwards annually up to 10 years
  Stratum 1 - randomisation related question was closed in December 2018; patients are in active follow-up: To show that a non total body irradiation (TBI) containing conditioning (Flu/Thio/ivBu or Flu/Thio/Treo) results in a non-inferior survival as compared to conditioning with TBI/Etoposide in children older than 4 years after HSCT from a Human leucocyte antigen (HLA) identical sibling donor (MSD) or a HLA matched donor (MD). The primary endpoint is the OS calculated from the date of the randomisation. Death from any cause will be considered an event.
Event free survival (EFS) Stratum 2 (mismatched donor transplantation) | first: 18 months after inclusion of first patient, afterwards annually up to 10 years
  EFS after allogeneic HSCT. EFS calculated from date of recruitment to disease progression or relapse, secondary neoplasm and death from any cause.
Overall Survival (OS), Stratum 1b: MSD/MD without randomisation | first: 18 months after inclusion of first patient, afterwards annually up to 10 years
  To explore the impact of risk factors on the incidence of adverse events of special interest (AESIs) and on overall survival and event free survival in the entire MSD/MD cohort

SECONDARY OUTCOMES:
EFS (Stratum 1a and 1b) | first: 18 months after inclusion of first patient, afterwards annually up to 10 years
  EFS calculated from date of randomization (1a) or recruitment (1b) to disease progression or relapse, secondary neoplasm and death from any cause. Patients lost to follow-up without event will be censored at the date of their last follow-up evaluation.
TRM | first: 18 months after inclusion of first patient, afterwards annually up to 10 years
  Cumulative Incidence of Treatment-related mortality (TRM) for Stratum 1 and 2.
Relapse/progression | first: 18 months after inclusion of first patient, afterwards annually up to 10 years
  Cumulative Incidence of Relapse for Stratum 1a, 1b and 2.
Acute and late toxicity for Stratum 1a, 1b and 2 | first: 18 months after inclusion of first patient, afterwards annually up to 10 years
  according a preselection out of CTC3
OS (Stratum 2) | first: 18 months after inclusion of first patient, afterwards annually up to 10 years
  The primary endpoint is the OS calculated from the date of the recruitment . Death from any cause will be considered an event.

OTHER OUTCOMES:
Acute Graft versus Host Disease (aGVHD) | first: 18 months after inclusion of first patient, afterwards annually up to 10 years
  According to the modified Seattle Glucksberg criteria
Secondary malignancies | first: 18 months after inclusion of first patient, afterwards annually up to 10 years
  Incidence, type and timepoint of occurence
Chronic Graft-versus-host disease (cGvHD) | first: 18 months after inclusion of first patient, afterwards annually up to 10 years
  Chronic GVHD is diagnosed using criteria created through the NIH consensus development project

CONTACTS AND LOCATIONS:
Overall Officials: Christina Peters, Prof. MD PhD, Study Chair — St. Anna Kinderspital, Vienna, Austria; Peter Bader, Prof. MD PhD, Study Chair — Goethe University; Franco Locatelli, Prof. MD PhD, Study Chair — Ospedale Pediatrico Bambino Gesù, Rome, Italy
Locations (119):
- Argentina (2):
  - Hospital de Pediatria "Juan P. Garrahan" Combate de Los Pozos N°1800 CABA, Buenos Aires
  - Hospital Sor Maria Ludovica, Department Hematology Stem Cell Transplant Unit, La Plata
- Australia (5):
  - Children's Cancer Centre The Royal Children's Hospital, Melbourne
  - Princess Margaret Hospital for Children, Perth
  - Sydney Children's Hospital, Randwick
  - Lady Cilento Children's Hospital, South Brisbane
  - The Children's Hospital at Westmead Oncology Unit, Sydney
- Austria (3):
  - Universitätsklinik für Kinder- und Jugendheilkunde, Abt. f. Hämato-Onkologie, Graz
  - Universitätsklinik für Kinder- und Jugendheilkunde, Innsbruck
  - St. Anna Children's Hospital, Vienna, Austria, Vienna
- Belarusian Research Center for Pediatric Oncology, Hematology and Immunology, Minsk, Belarus
- Belgium (5):
  - Hôpital Universitaire des Enfants Reine Fabiola (HUDERF), Brussels
  - Cliniques Universitaires Saint-Luc (UCL) Hématologie et oncologie pédiatrique, Brussels
  - University Hospital Gent Pediatrische hemato-oncologie, Ghent
  - University Hospitals Leuven Kinderhemato-oncologie, Leuven
  - Centre Hospitalier Universitaire de Liège Domaine Universitaire du Sart Tilman, Liège
- Canada (6):
  - Alberta Children's Hospital Division of Pediatric Oncology, Calgary
  - Montreal Children's Hospital, Montral
  - CHU Sainte-Justine Hematology-Oncology Division, Montreal
  - Hospital for Sick Children University of Toronto Division of Haematology/Oncology, Toronto
  - BC Children's Hospital, Vancouver
  - CancerCare Manitoba/University of Manitoba, Winnipeg
- Hospital Dr Luis Calvo Mackenna, Santiago, Chile
- Department of Pediatrics, UHC Zagreb, Zagreb, Croatia
- Department of Pediatric Hematology and Oncology Teaching Hospital Motol, 2nd Medical School, Charles University, Prague, Czechia
- Paediatric Stem Cell Transplant and Immune Deficiency, Dept. for children and adolescents 4072, Rigshospitalet, Copenhagen, Denmark
- Division of Hematology-Oncology and Stem Cell Transplantation, Hospital for Children and Adolescents, Univ. of Helsinki, Helsinki, Finland
- France (13):
  - CHU Bordeaux, Bordeaux
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble - Clinique Universitaire de Pédiatrie, Hôpital Couple Enfant, Grenoble
  - CHRU Lille, Service d'Hématologie Pédiatrique, Lille
  - IHOP / Lyon, Service Hématologie et d'Oncologie pédiatrique, Lyon
  - Hopital la Timone Adulte, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - CHU Nancy - Hopital d'Enfants, Nancy
  - CHU Nantes, Service d'onco hémato pédiatrie, Nantes
  - Hôpital Robert Debré, Paris
  - CHU de Rennes, Serive d'Onco-Pédiatrie, Rennes
  - CHU de Rouen, Hopital des Enfants, Service d' Immuno-Hématologie Oncologie Pédiatrique, Rouen
  - CHU Strasbourg, Service d'hématologie et d'oncologie pédiatrique, Strasbourg
- Germany (24):
  - Uniklinik RWTH Aachen, Kinder- und Jugendmedizin, Aachen
  - Charité - Universitätsmedizin Berlin, Campus Virchow-Klinikum, Berlin
  - Universitätsklinikum Bonn, Abteilung für Pädiatrische Hämatologie und Onkologie, Bonn
  - Universitätsklinikum Düsseldorf, Klinik für Kinder-Onkologie, -Hämatologie und Klinische Immunologie, Düsseldorf
  - Universitätsklinikum Erlangen, Kinder- und Jugendklinik, Erlangen
  - Universitätsklinikum Essen, Klinik für Kinderheilkunde III, Essen
  - Klinikum der Johann Wolfgang Goethe-Universität, Klinik für Kinder- und Jugendmedizin (KKJM), Frankfurt am Main
  - Universitätsklinikum Freiburg, Zentrum für Kinder- und Jugendmedizin, Freiburg im Breisgau
  - Universitätsklinikum Gießen, Zentrum für Kinder- und Jugendmedizin, Giessen
  - Universitätsmedizin Greifswald, Klinik und Poliklinik für Kinder- und Jugendmedizin, Greifswald
  - Universitätsklinikum Halle (Saale), Universitätsklinik und Poliklinik für Kinder- und Jugendmedizin, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Klinik und Poliklinik für Pädiatrische Hämatologie und Onkologie, Hamburg
  - Medizinische Hochschule Hannover, Zentrum Kinderheilkunde und Jugendmedizin, Hanover
  - Universitätsklinikum Heidelberg, Zentrum für Kinder- und Jugendmedizin, Heidelberg
  - Universitätsklinikum Jena, Sektion für Stammzelltransplantation, Jena
  - UKSH - Universitätsklinikum Schleswig-Holstein, Klinik für Allgemeine Pädiatrie, Kiel
  - Universitätsmedizin Leipzig, Abteilung für Pädiatrische Onkologie, Hämatologie und Hämostaseologie, Leipzig
  - Klinikum der Universität München, Dr. von Haunersches Kinderspital, München
  - Städt. Krankenhaus München Schwabing, Universitätskinderklinik der TU München, München
  - Universitätsklinikum Münster, Klinik für Kinder- und Jugendmedizin, Münster
  - Universitätsklinikum Regensburg, Klinik und Poliklinik für Kinder- und Jugendmedizin, Regensburg
  - Universitätsklinik für Kinder- und Jugendmedizin Tübingen, Tübingen
  - Universitätsklinikum Ulm, Klinik für Kinder- und Jugendmedizin, Ulm
  - Universitäts-Kinderklinik Würzburg, Würzburg
- Saint Sophia Children's Hospital BMT Unit, Athens, Greece
- National Institute of Haematology and Infectious Disease, Hospital of Southern Pest, Paediatric Bone Marrow Transplantation Unit, Budapest, Hungary
- Israel (3):
  - Rambam Medical Center, Haifa
  - Schneider Children's Medical Center of Israel, Petah Tikva
  - Dana Children's Hospital, Tel Aviv
- Italy (10):
  - Azienda Ospedaliero-Universitaria Policlinico S. Orsola-Malpighi di Bologna, Bologna
  - Ospedale Mayer di Firenze SODc Tumori Pediatrici e TMO, Florence
  - Istituto Gaslini Genova Oncoematologia Pediatrica-, Genoa
  - A.O. San Gerardo di Monza Clinica Pediatrica, Monza
  - A.O.R.N. Santobono Pausilipon, Dipartimento di Oncoematologia, Napoli
  - Azienda Ospedaliera di Padova Oncoematologia Pediatrica, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana U.O. di Oncoematologia Pediatrica A.O., Pisa
  - Ospedale Pediatrico Bambino Gesù, Sapienza, University of Rome, Rome
  - Ospedale Infantile Regina Margherita SC Oncoematologia e Centro Trapianti, Torino
- University of Malaya, Department of Paediatrics, Kuala Lumpur, Malaysia
- Instituto Nacional de Peditria, Mexico City, Mexico
- Netherlands (2):
  - Leiden University Medical Center Department of Pediatrics/BMT unit, Leiden
  - Princess Máxima Center for Pediatric Oncology, Utrecht
- Starship Children's Hospital, Auckland, New Zealand
- Oslo University Hospital Rikshospitalet, Oslo, Norway
- Poland (5):
  - University Hospital No.1, Collegium Medicum UMK, department of Paediatrics, Oncology, Hematology and Paediatric Transplantology, Bydgoszcz
  - University Children's Hospital in Krakow, Department of Transplantation, Krakow
  - Children's University Hospital, Dept. Pediatric Hematology, Oncology, and Transplantology, Lublin
  - Poznan University of Medical Sciences, Department of Pediatric Onology, Hematology & HSCT, Poznan
  - Cape of Hope, Wroclaw Medical University, Wroclaw
- Romania (2):
  - IInsitutul Clinic Fundeni, Sectia de Transplant Medular, Bucharest
  - University of Medicine and Pharmacy V. BABES, Emergency Children's Hospital LOUIS TURCANU, III. Clinic of Pediatrics , Department of Onco-hematology and Bone Marrow Transplantation, Timișoara
- King Abdullah specialists children hospital, Riyadh, Saudi Arabia
- University Children's Hospital, Bratislava, Slovakia
- University childrens' hospital, UMCL, Ljubljana, Slovenia
- Spain (5):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Materno Infantil de Málaga, Málaga
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
- Sweden (4):
  - Queen Silvia Children's Hospital, Department of Pediatric Oncology (Avdelnig 321-322), Gothenburg
  - Skane University Hospital, Dept. of Pediatrics, Section for Hematology and Oncology, Lund
  - Karolinska University Hospital, Department of Pediatrics, Stockholm
  - University Children's Hospital, Dept. of Women's & Children's Health Section for Pediatrics, Uppsala
- Switzerland (3):
  - Universitäts-Kinderspital beider Basel (UKBB), Basel
  - HUG Hôpitaux Universitaire de Genève, Geneva
  - Universitäts-Kinderspital Zurich, Zurich
- Turkey (Türkiye) (12):
  - Ankara University School of Medicine Pediatric Stem Cell Transplantation Unit, Ankara
  - Gazi University School of Medicine Pediatric Stem Cell Transplantation Unit, Ankara
  - Gülhane Training and Research Hospital, Ankara
  - Akdeniz University School of Medicine Pediatric Stem Cell Transplantation Unit, Antalya
  - Bahcesehir University School of Medicine Pediatric Stem Cell Transplantation Unit, Antalya
  - Acibadem University Atakent Hospital Pediatric Stem Cell Transplantation Unit, Istanbul
  - Bahcelievler Medicalpark Hospital Pediatric Stem Cell Transplantation Unit, Istanbul
  - Bahcesehir University School of Medicine Pediatric Stem Cell Transplantation Unit, Istanbul
  - Medipol Mega Üniversite Hastanesi, Istanbul
  - Dokuzeylul University School of Medicine Pediatric Stem Cell Transplantation Unit, Izmir
  - Ege University School of Medicine Pediatric Stem Cell Transplantation Unit, Izmir
  - Erciyes University School of Medicine Pediatric Stem Cell Transplantation Unit, Kayseri

REFERENCES:
- [Derived] Buechner J, Poetschger U, Bader P, Yesilipek MA, Pichler H, Palma J, Staciuk R, Riha P, Krivan G, Ifversen M, Gungor T, Goussetis E, Kalwak K, Toporski J, Gabriel M, Renard MM, Diaz-de-Heredia C, Matic T, Calkoen FG, Svec P, Meisel R, Balduzzi AC, Locatelli F, Peters C, Dalle JH, Stein J. Outcome of children with B-cell acute lymphoblastic leukemia with hypodiploidy or BCR::ABL1 fusion undergoing allogeneic HSCT. Blood. 2025 Nov 19:blood.2025030951. doi: 10.1182/blood.2025030951. Online ahead of print. PMID 41259231
- [Derived] Kalwak K, Moser LM, Potschger U, Bader P, Kleinschmidt K, Meisel R, Dalle JH, Yesilipek A, Balduzzi A, Krivan G, Goussetis E, Staciuk R, Sedlacek P, Pichler H, Svec P, Gabriel M, Gungor T, Bilic E, Buechner J, Renard M, Vettenranta K, Ifversen M, Diaz-de-Heredia C, Stein J, Toporski J, Bierings M, Peters C, Ansari M, Locatelli F. Comparable outcomes after busulfan- or treosulfan-based conditioning for allo-HSCT in children with ALL: results of FORUM. Blood Adv. 2025 Feb 25;9(4):741-751. doi: 10.1182/bloodadvances.2024014548. PMID 39602342
- [Derived] Bader P, Potschger U, Dalle JH, Moser LM, Balduzzi A, Ansari M, Buechner J, Gungor T, Ifversen M, Krivan G, Pichler H, Renard M, Staciuk R, Sedlacek P, Stein J, Heusel JR, Truong T, Wachowiak J, Yesilipek A, Locatelli F, Peters C. Low rate of nonrelapse mortality in under-4-year-olds with ALL given chemotherapeutic conditioning for HSCT: a phase 3 FORUM study. Blood Adv. 2024 Jan 23;8(2):416-428. doi: 10.1182/bloodadvances.2023010591. PMID 37738088
- [Derived] Gomez SM, Varela MA, Ruiz C, Sung L. Comparable Outcomes of Matched Sibling Donor and Matched Unrelated Donor Stem Cell Transplantation in Children With Acute Leukemia in Argentina. J Pediatr Hematol Oncol. 2021 Oct 1;43(7):e1020-e1024. doi: 10.1097/MPH.0000000000002174. PMID 33974585
- [Derived] Peters C, Dalle JH, Locatelli F, Poetschger U, Sedlacek P, Buechner J, Shaw PJ, Staciuk R, Ifversen M, Pichler H, Vettenranta K, Svec P, Aleinikova O, Stein J, Gungor T, Toporski J, Truong TH, Diaz-de-Heredia C, Bierings M, Ariffin H, Essa M, Burkhardt B, Schultz K, Meisel R, Lankester A, Ansari M, Schrappe M; IBFM Study Group;; von Stackelberg A; IntReALL Study Group; Balduzzi A; I-BFM SCT Study Group; Corbacioglu S; EBMT Paediatric Diseases Working Party; Bader P. Total Body Irradiation or Chemotherapy Conditioning in Childhood ALL: A Multinational, Randomized, Noninferiority Phase III Study. J Clin Oncol. 2021 Feb 1;39(4):295-307. doi: 10.1200/JCO.20.02529. Epub 2020 Dec 17. PMID 33332189
- [Derived] Tasian SK, Peters C. Targeted therapy or transplantation for paediatric ABL-class Ph-like acute lymphocytic leukaemia? Lancet Haematol. 2020 Dec;7(12):e858-e859. doi: 10.1016/S2352-3026(20)30369-0. No abstract available. PMID 33242441
- [Derived] Choong E, Uppugunduri CRS, Marino D, Kuntzinger M, Doffey-Lazeyras F, Lo Piccolo R, Chalandon Y, Peters C, Daali Y, Ansari M. Therapeutic Drug Monitoring of Busulfan for the Management of Pediatric Patients: Cross-Validation of Methods and Long-Term Performance. Ther Drug Monit. 2018 Feb;40(1):84-92. doi: 10.1097/FTD.0000000000000468. PMID 29189665
- See also: St. Anna Kinderkrebsforschung — https://kinderkrebsforschung.at/
- See also: St. Anna Kinderspital — https://www.stanna.at/
- See also: Peters C et al. Total Body Irradiation or Chemotherapy Conditioning in Childhood ALL: A Multinational, Randomized, Noninferiority Phase III Study. J Clin Oncol. 2021 Feb 1;39(4):295-307 — https://pubmed.ncbi.nlm.nih.gov/33332189/